CLINICAL TRIAL: NCT04429516
Title: PAciFy Cough: A Multicentre, Double Blind, Placebo Controlled, Crossover Trial of Morphine Sulfate for the Treatment of PulmonAry Fibrosis Cough
Brief Title: Morphine Sulfate/Placebo for the Treatment of PulmonAry Fibrosis Cough
Acronym: PAciFy Cough
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RBH2019/001; 2019-003571-19 (EudraCT Number)
Record Dates: First submitted 2020-03-12; First posted 2020-06-12 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine Sulfate (Experimental)
  Interventions: Drug: Morphine Sulfate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Morphine Sulfate — over-encapsulated Morphine Sulfate prolonged release 5mg tablet, twice daily for 14 days. Patients will then crossover after a 7 day wash out period.
  Arms: Morphine Sulfate
Drug: Placebo oral tablet — capsule containing Microcrystalline Cellulose Ph. Eur, 5 mg twice daily
  Arms: Placebo

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a disease of unknown cause that results in scarring of the lungs.

Cough is reported by 85% of patients with IPF and can be a distressing symptom with significant physical, social and psychological consequences particularly anxiety and depression.

The cause of cough in IPF is poorly understood and there are currently no proven effective therapies. Morphine has long been advocated for the suppression of chronic cough in other conditions. While morphine is frequently used as a palliative agent for breathlessness in IPF, its effects on cough have never been tested. The aim of this study is therefore to explore and compare the effect of low dose morphine, one of the few therapies shown to be effective in some patients with otherwise refractory chronic cough, in patients with IPF, to an inactive substance known as a placebo.

To make a fair comparison, patients will be randomly allocated to receiving either morphine or placebo in a blinded fashion. This means neither the doctor nor the patient will know which drug they are receiving, and the drugs will appear the same. However, the trial is designed so that you will receive both morphine and placebo, but at different times (this is called a cross-over study). More specifically, you will be given either morphine or placebo for 14 days at a time.

In this study, it is hypothesised that compared with placebo, low dose (5mg) controlled release Morphine sulfate (MST) will reduce the number of coughs recorded during a 24hr period in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported cough (> 8 weeks), with cough VAS ≥ 30/100
2. A diagnosis of IPF within 5 years prior to the screening visit, as per applicable ATS/ERS/JRS/ALAT guidelines, in line with hospital records.
3. Age 3.1. Male and female participants aged ≥ 40 - 90 years at the time of signing informed consent
4. Sex:

   4.1 Male participants: A male participant must agree to use contraception as detailed in Appendix 2 of this protocol during the study and for at least 90 days after the follow-up visit, and refrain from donating sperm during this period 4.2 Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP)
5. Meeting all of the following criteria during the screening period: FVC ≥ 45% predicted of normal, Forced expiratory volume in 1 second (FEV1)/FVC ≥0.7, DLCO corrected for Hb ≥30% predicted of normal.
6. The extent of fibrotic changes is greater than the extent of emphysema on the most recent HRCT scan (investigator determined within 24 months of the study screening visit)
7. Written informed consent.

Exclusion criteria:

1. Treatment with immunosuppressive therapy or antibiotics within last 4 weeks. A stable dose of corticosteroids equivalent to prednisolone of 10 mg per day or less, if used for an indication other than pulmonary disease will be permitted
2. Current smoker
3. History of alcohol and drug(s) addiction
4. Regular use of sedative therapies
5. Acute IPF exacerbation within 6 months prior to screening and/or during the screening period.
6. Concurrent use of pirfenidone or Nintedanib, unless receiving a stable dose for at least 8 weeks prior to screening
7. Use of ACE inhibitors
8. Patients with co-existent conditions know to be associated with the development of fibrotic lung disease. This includes: connective tissue disease, (plural plaques, mesothelioma), granulomatous disease including sarcoidosis. Patient with auto-immune profile considered diagnostic for a specific connective tissue disease will be excluded, even in the absence of systemic symptoms. Non-specific rises in auto antibodies e.g. rheumatoid factors, anti-nuclear antibody etc. will not be used to exclude individuals from the study.
9. Significant other organ co-morbidity including hepatic or renal impairment and pulmonary hypertension (investigator determined).
10. Significant coronary artery disease (myocardial infarction within 6 months or ongoing unstable angina within 4 weeks of screening visit) or congestive cardiac failure based on clinical examination
11. Patients as significant risk of side effects, intolerance or allergy to morphine
12. Pregnant and breastfeeding patients, or women or child-bearing potential, not using a reliable contraceptive method (see Appendix 2). A urine pregnancy test will be performed in females of child-bearing potential at the initial study visit.
13. Unable to provide informed written consent
14. Predicted life expectancy < 6 months
15. Use of long-term oxygen therapy. Use of ambulatory oxygen will be permitted.
16. Current or use of opiates within 14 days of the screening visit.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
The percent change in daytime cough frequency (coughs per hour) | from baseline as assessed by objective digital cough monitoring at Day 14 of treatment

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life scores (Living with Idiopathic Pulmonary Fibrosis Questionnaire) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  Living with Idiopathic Pulmonary Fibrosis (L-IPF): Developing a Patient-Reported Symptom and Impact Questionnaire to Assess Health-Related Quality of Life in IPF; on a scale between 0 to 4, where 0 is Not at all and 4 is Extremlly.
Change from baseline in health-related quality of life scores (HDAS- Hospital Anxiety and Depression Scale) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  HADS - Hospital Anxiety and Depression Scale (Scoring 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case).
Change from baseline in health-related quality of life scores (K-BILD - King's Brief Interstitial Lung Disease Questionnaire) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  The KBILD is a self-completed health status questionnaire that comprises 15 items and a seven-point Likert response scale. It has three domains: psychological, breathlessness and activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 represents best health status.
Change from baseline in self-reported cough (Leicester Cough Questionnaire (LCQ) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  The Leicester Cough Questionnaire comprises of 19 questions, each on a score between 1 to 7, the latter meaning worse outcome. 8 of the questions assess the physical cough domain, 7 items assess the psychological impact of cough, and 4 questions assess the social impact of cough.
Change from baseline in self-reported cough - Visual analogue scale (VAS) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  VAS - The cough visual analogue scale (VAS) represents a simple instrument, using a 100 mm linear scale where patient can indicate the severity of their cough between the two extremes: zero is no cough while 100 mm is the worst cough imaginable.
Change from baseline in Dyspnoea (Dyspnoea 12) | At Day 0, Day 14, Day 22, Day 36 and Day 50-64
  D-12 consists of 12 descriptor items on a scale of none (0), mild (1), moderate (2), or severe (3). It provides an overall score for breathlessness severity that incorporates seven physical items and five affective items
Change from baseline in global impression of change in quality of life, cough and breathlessness. | At Day 14 and Day 36
  It provides a brief, stand-alone assessment of treatment effect on cough, breathlessness and overall quality of live on a scale of: worse, same and better.
Proportion of responders with a minimum of 20% decrease from baseline at the end of treatment in 24-hour average cough count. | Comparison made between pre-treatment and at follow up visit in both the first and then the crossover arms of the study: Day 0, Day 14, Day 22 and Day 36

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hope-Gill BD, Hilldrup S, Davies C, Newton RP, Harrison NK. A study of the cough reflex in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2003 Oct 15;168(8):995-1002. doi: 10.1164/rccm.200304-597OC. Epub 2003 Aug 13. PMID 12917229
- [Background] van Manen MJ, Birring SS, Vancheri C, Cottin V, Renzoni EA, Russell AM, Wijsenbeek MS. Cough in idiopathic pulmonary fibrosis. Eur Respir Rev. 2016 Sep;25(141):278-86. doi: 10.1183/16000617.0090-2015. PMID 27581827
- [Background] Morice AH, Menon MS, Mulrennan SA, Everett CF, Wright C, Jackson J, Thompson R. Opiate therapy in chronic cough. Am J Respir Crit Care Med. 2007 Feb 15;175(4):312-5. doi: 10.1164/rccm.200607-892OC. Epub 2006 Nov 22. PMID 17122382
- [Background] Bajwah S, Davies JM, Tanash H, Currow DC, Oluyase AO, Ekstrom M. Safety of benzodiazepines and opioids in interstitial lung disease: a national prospective study. Eur Respir J. 2018 Dec 6;52(6):1801278. doi: 10.1183/13993003.01278-2018. Print 2018 Dec. PMID 30309973
- [Derived] Wu Z, Spencer LG, Banya W, Westoby J, Tudor VA, Rivera-Ortega P, Chaudhuri N, Jakupovic I, Patel B, Thillai M, West A, Wijsenbeek M, Maher TM, Smith JA, Molyneaux PL. Morphine for treatment of cough in idiopathic pulmonary fibrosis (PACIFY COUGH): a prospective, multicentre, randomised, double-blind, placebo-controlled, two-way crossover trial. Lancet Respir Med. 2024 Apr;12(4):273-280. doi: 10.1016/S2213-2600(23)00432-0. Epub 2024 Jan 15. PMID 38237620
- [Derived] Wu Z, Banya W, Chaudhuri N, Jakupovic I, Maher TM, Patel B, Spencer LG, Thillai M, West A, Westoby J, Wijsenbeek M, Smith J, Molyneaux PL. PAciFy Cough-a multicentre, double-blind, placebo-controlled, crossover trial of morphine sulphate for the treatment of pulmonary Fibrosis Cough. Trials. 2022 Mar 2;23(1):184. doi: 10.1186/s13063-022-06068-4. PMID 35236391